CLINICAL TRIAL: NCT01176500
Title: A Pilot, Open-Label, Proof-of-Concept Study of the Use of [18F]Fluciclatide PET/CT Imaging in the Evaluation of Anti-Angiogenic Therapy in Solid Tumors
Brief Title: A Pilot, Open-label Study of 18F-Fluciclatide PET/CT Imaging in the Evaluation of Anti-angiogenic Therapy in Solid Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH); GE Healthcare (Industry)
Responsible Party: Karen A. Kurdziel, M.D./NIH Clinical Center, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 100173; 10-C-0173
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-11-18

CONDITIONS: Colon Cancer; Lung Cancer; Cervical Cancer; Renal Cell Carcinoma; Uterine Cancer
Keywords: PET Imaging; (18F)Fluciclatide; Anti-Angiogenic Therapies; Solid Tumors
MeSH Terms: conditions — Colonic Neoplasms; Lung Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Renal Cell; Uterine Neoplasms

INTERVENTIONS:
Drug: (18)Fluciclatide

SUMMARY:
Background:

* Fluciclatide is a small cyclic peptide containing the RGD tri-peptide, which preferentially binds with high affinity to alpha(v)beta(3) integrins, which are up-regulated in and may regulate angiogenesis.
* [18F]Fluciclatide is a new radiopharmaceutical developed for PET imaging
* Changes in [18F]fluciclatide uptake will be evaluated before and after treatment of patients with targeted antiangiogenic drugs

Objectives:

Primary

* To determine tumor uptake and retention of [18F]fluciclatide before and after 1 cycle of treatment with targeted anti-angiogenic therapy
* Secondary
* To assess the safety of multiple intravenous (IV) administrations of Fluciclatide [18F] Injection in subjects with solid tumors
* To obtain preliminary data on the relationships between [18F]fluciclatide as a pharmacodynamic marker and standard of care imaging markers of clinical response (e.g. contrast-enhanced (CE) static computed tomography (CT), bone scintigraphy, FDG-PET), obtained as part of routine clinical follow-up as specified in the referring protocols, as well as any optional imaging performed

Eligibility:

* Patients greater than or equal to 18 years, with documented malignancy, and solid tumor greater than or equal to 1 cm outside of the liver, who are scheduled to enroll in an NCI therapy protocol using one of the anti-angiogenic agents described in the full protocol
* Platelet count greater than 75,000 x 10(6)/L, hemoglobin greater than 9g/dL, prothrombin time (PT) and aPTT less than 2 times normal limits.
* The subject has not received any targeted anti-angiogenic agents within 60 days prior to pre-treatment (baseline) [18F]fluciclatide administration

Design:

This study is intended to obtain preliminary data on the uptake and retention of [18F]fluciclatide before and after anti-angiogenic therapy. This will enable optimization of the imaging protocol, identification of the most relevant imaging parameters, and allow for calculation of the number patients required to power a larger study to assess the utility of PET imaging with [18F]fluciclatide as a pharmacodynamic biomarker in the context of targeted anti-angiogenic therapies. We expect to enroll 30 evaluable patients in this single center study. Subjects will undergo at least two [18F]fluciclatide PET/CT imaging studies, one pre-therapy and one following completion of 1 cycle of chemotherapy. An optional early post-therapy (2-7 days post therapy commencement) [18F]fluciclatide PET/CT may be performed. The magnitude of [18F]fluciclatide uptake on the pre- and post- treatment PET/CT studies will be evaluated to determine if there is a measureable difference in uptake. Data from the subject's referring therapy protocol will be reviewed for up to one year. An optional DCE-MRI scans of the target lesion may also be performed.

DETAILED DESCRIPTION:
Background:

* Fluciclatide is a small cyclic peptide containing the RGD tri-peptide, which preferentially binds with high affinity to alpha(v)beta(3) integrins, which are up-regulated in and may regulate angiogenesis.
* [18F]Fluciclatide is a new radiopharmaceutical developed for PET imaging
* Changes in [18F]fluciclatide uptake will be evaluated before and after treatment of patients with targeted antiangiogenic drugs

Objectives:

Primary

* To determine tumor uptake and retention of [18F]fluciclatide before and after 1 cycle of treatment with targeted anti-angiogenic therapy
* Secondary
* To assess the safety of multiple intravenous (IV) administrations of Fluciclatide [18F] Injection in subjects with solid tumors
* To obtain preliminary data on the relationships between [18F]fluciclatide as a pharmacodynamic marker and standard of care imaging markers of clinical response (e.g. contrast-enhanced (CE) static computed tomography (CT), bone scintigraphy, FDG-PET), obtained as part of routine clinical follow-up as specified in the referring protocols, as well as any optional imaging performed

Eligibility:

* Patients greater than or equal to 18 years, with documented malignancy, and solid tumor greater than or equal to 1 cm outside of the liver, who are scheduled to enroll in an NCI therapy protocol using one of the anti-angiogenic agents described in the full protocol
* Platelet count greater than 150,000 x 10(6)/L, hemoglobin greater than 9g/dL, prothrombin time (PT) and aPTT less than 2 times normal limits.
* The subject has not received any targeted anti-angiogenic agents within 60 days prior to pre-treatment (baseline) [18F]fluciclatide administration

Design:

This study is intended to obtain preliminary data on the uptake and retention of [18F]fluciclatide before and after anti-angiogenic therapy. This will enable optimization of the imaging protocol, identification of the most relevant imaging parameters, and allow for calculation of the number patients required to power a larger study to assess the utility of PET imaging with [18F]fluciclatide as a pharmacodynamic biomarker in the context of targeted anti-angiogenic therapies. We expect to enroll 30 evaluable patients in this single center study. Subjects will undergo at least two [18F]fluciclatide PET/CT imaging studies, one pre-therapy and one following completion of 1 cycle of chemotherapy. An optional early post-therapy (2-7 days post therapy commencement) [18F]fluciclatide PET/CT may be performed. The magnitude of [18F]fluciclatide uptake on the pre- and post- treatment PET/CT studies will be evaluated to determine if there is a measureable difference in uptake. Data from the subject's referring therapy protocol will be reviewed for up to one year. An optional DCE-MRI scans of the target lesion may also be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult subjects (greater than or equal to18 years old), with documented malignancy, with at least one solid tumor greater than or equal to 1 cm in diameter (not within the liver), who are scheduled to enroll in an NCI therapy protocol using one of the anti-angiogenic therapy agents (Vandetanib, Cediranib or Bevacizumab)
* The subject has a platelet count of 150,000 x 10(6)/L, hemoglobin value of greater than 9 g/dL, PT and an aPTT less than 2 times normal limits.
* The subject has a clinically acceptable medical history, physical examination and vital signs findings during the screening period (from less than 4 weeks before administration of Fluciclatide (18F) Injection); i.e. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2.
* The subject has had no open surgical wounds in close proximity to the target lesion(s) within 10 days prior to study entry.
* The subject has not had a biopsy of the target lesion within 7 days of PET/CT imaging.
* The subject has not had radiation therapy to the region of the target lesion.
* Enrolling in the following NCI anti-angiogenic therapy protocols:

  08-C-0020

  09-C-0192

  07-C-0058

  09-C-0019

EXCLUSION CRITERIA:

* The subject is pregnant or lactating.
* The subject is being treated with doses of heparin or warfarin resulting in elevation of PT or aPTT greater than 2 times normal.
* The subject has received any anti-angiogenic agent (e.g. bevacizumab, sorafenib, sunitinib) within 60 days prior to pre-treatment (baseline) [18F]fluciclatide PET imaging. This stipulation does not apply after the baseline [18F]fluciclatide PET imaging.
* The subject has received another investigational medicinal product (IMP) within 24 hours before or is scheduled to receive another IMP within 24 hours after Fluciclatide (18F) Injection.
* The subject has any contraindication to any of the study procedures, products used or its constituents (e.g. severe claustrophobia unrelieved by oral anxiolytics).
* The subject is unable to lie still for 75 minutes.
* The subject is known to have a history of hyper- or hypo-coagulation syndromes resulting in prolongation of bleeding parameters. Such coagulopathies include but are not limited to Von Willebrand disease, Protein C deficiency, Protein S deficiency, Hemophilia A/B/C, Factor-V Leiden, and Bernard-Soulier syndrome.
* The subject has undergone a surgical procedure to the target lesion within 28 days prior to baseline [18F]fluciclatide administration OR is scheduled to undergo a surgical procedure between the baseline and post 1-cycle [18F]fluciclatide PET/CT.
* The subject has only bone metastasis

ADDITIONAL INCLUSION CRITERIA FOR SUBJECTS UNDERGOING OPTIONAL MR:

-Serum creatinine within 2 weeks prior to MRI less than or equal to 1.8mg/dl and estimated glomerular filtration rate (eGFR) must be greater than 30 ml/min/1.73m(2).

ADDITIONAL EXCLUSION CRITERIA FOR SUBJECTS UNDERGOING OPTIONAL MR:

* The subject has known allergy to gadolinium
* The subject has contraindications to MRI:

  * Subjects must weigh less than 136 kg (weight limit for scanner table).
  * Subjects cannot have pacemakers, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices or metal not compatible with MRI.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07-28; Primary Completion 2011-11-18 (Actual); Study Completion 2011-11-18 (Actual)

PRIMARY OUTCOMES:
To determine tumor uptake and retention of [18F]fluciclatide before and after 1 cycle of treatment with targeted anti-angiogenic therapy. | 2 years

SECONDARY OUTCOMES:
To obtain preliminary data on the relationships between [18F]fluciclatide as a pharmacodynamic marker and standard of care imaging markers of clinical response. | 2 years
To assess the safety of multiple intravenous (IV) administrations of Fluciclatide [18F] Injection in subjects with solid tumors. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brooks PC, Clark RA, Cheresh DA. Requirement of vascular integrin alpha v beta 3 for angiogenesis. Science. 1994 Apr 22;264(5158):569-71. doi: 10.1126/science.7512751.
- [Background] Line BR, Mitra A, Nan A, Ghandehari H. Targeting tumor angiogenesis: comparison of peptide and polymer-peptide conjugates. J Nucl Med. 2005 Sep;46(9):1552-60. PMID 16157540
- [Background] Egeblad M, Werb Z. New functions for the matrix metalloproteinases in cancer progression. Nat Rev Cancer. 2002 Mar;2(3):161-74. doi: 10.1038/nrc745. PMID 11990853